CLINICAL TRIAL: NCT05350410
Title: A Pilot Study for the Healthy Actions and Lifestyles to Avoid Dementia or Hispanos y el ALTo a la Demencia Program (HALT-AD)
Brief Title: "Healthy Actions and Lifestyles to Avoid Dementia or Hispanos y el ALTo a la Demencia Program"
Acronym: HALT-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HALT-AD
Record Dates: First submitted 2022-04-06; First posted 2022-04-28 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-07

CONDITIONS: Dementia; Alzheimer's Disease; Dementia Prevention
Keywords: dementia; prevention; education; lifestyle modification; digital health
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This pilot study will be a longitudinal study of an inception cohort exposed to the HALT AD online educational program for a four month study. It will utilize pre- and post- intervention collection of quantitative and qualitative data to evaluate the program's first prototype. Cognitively normal midlife and older-adult participants will be eligible to participate in this pilot study with the following inclusion criteria:
  * Ages 50-85
  * Montreal Cognitive Assessment-Telephone/Blind version (T-MoCA) Score equal to or greater than 18/22
  * Sufficient proficiency in English or Spanish to undergo clinical assessment and participate
  * Technical ability to participate
  * Sufficient vision and hearing to participate 20 participants will be enrolled at UCSD
  * 10 will complete the English version
  * 10 will complete the Spanish version
  Aim to recruit 50% women and enroll a diverse participant sample across varied age ranges within both language groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HALT-AD (Experimental): HALT-AD is an online educational program designed to teach about dementia and lifestyle changes that can help preserve brain health and lower dementia risk. Participants complete online courses and engage in facilitated discussion groups.
  Interventions: Behavioral: HALT-AD

INTERVENTIONS:
Behavioral: HALT-AD — HALT-AD is an online educational program designed to teach about dementia and lifestyle changes that can help preserve brain health and lower dementia risk. Participants complete online courses and engage in facilitated discussion groups.

SUMMARY:
A Pilot Study for the Healthy Actions and Lifestyles to Avoid Dementia or Hispanos y el ALTo a la Demencia program (HALT-AD). This initial four-months pilot study will focus on at least three educational courses (introduction to dementia and lifestyle risk factors, sleep and diet). It may also include a fourth educational course on social connectivity and loneliness. Completion of this initial pilot study will allow for a round of improvements informed by data from the program, on usability, as well as feedback from participants and citizen advisors. This will allow for an iterative process to build the program to its full content, with feedback to optimize the user experience and ensure the accessibility of the content. The information generated from this study will help inform the development of the second program's prototype, expected to benefit from the initial pilot to become more user-friendly, effective and accessible to the target audience.

This pilot study will be a longitudinal study of an inception cohort exposed to the HALT-AD online educational program for a four-month study. It will utilize pre- and post- intervention collection of quantitative and qualitative data to evaluate the program's first prototype.

DETAILED DESCRIPTION:
Healthy Actions and Lifestyles to Avoid Dementia or Hispanos y el ALTo a la Demencia program (HALT- AD) is a novel bilingual educational program that will focus on reducing risk factors with the ultimate goal of preventing dementia. It will be centered around a web-based interactive virtual online platform that will be developed to be dynamic, engaging, and interactive. Through interactive courses, the educational content of HALT-AD will provide guidance on modifiable lifestyle risk factors and the identification of treatable medical conditions including cerebrovascular health, sleep, sensory loss, social isolation, mood, diet, and physical activity.

Participants in HALT-AD will be provided with personalized risk profiles, will be encouraged to learn about risk factors and how they can effectively modify them, and will be provided with feedback on their progress. Participants will participate in facilitated support discussion groups, which will focus on the content of the educational material and the invocation of change through participant engagement and compliance.

Prior to launching the full HALT-AD program, it is essential that the Sponsor conduct a preliminary pilot study to evaluate the program's first prototype. At the end of the 3-month pilot program, evaluations will include: the usability of- and engagement with- the online platform and users' acceptability of the learning content and facilitated support discussion groups. As well as evaluating preliminary evidence on the effectiveness of the program in changing knowledge, self-efficacy, and dementia-related lifestyle risk factors. The program will also be evaluated on metrics such as being user friendly, engaging, supportive and communicative, with the potential for scalability to state- and national-levels.

Aims:

1. To evaluate engagement with- the online platform
2. To evaluate preliminary evidence on the effectiveness of the program in changing

   a) knowledge, b) self-efficacy, and c) dementia-related lifestyle risk factors
3. To determine users' acceptability of the program content
4. To determine users' acceptability and satisfaction with the facilitated support discussion groups
5. To evaluate the usability of the online platform

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained and documented (from the participant).
2. Sufficient proficiency in English or Spanish to undergo clinical assessment and participate in an online educational program.
3. Ages 50-85
4. Montreal Cognitive Assessment-Telephone/Blind Version (T-MoCA) score ≥18/22
5. Technical ability to participate in an online educational program (i.e. ability to operate a computer/tablet and gain internet access; ability to send and receive emails)
6. Sufficient vision and hearing to participate in online educational program (judgement of site investigator)
7. Ability to sit comfortably for a period of at least 30 minutes

Exclusion Criteria:

1. Participants who, in the opinion of the co-PIs, are not able to complete trial procedures or adhere to the schedule of study assessments will be excluded from study participation.
2. Individuals where English or Spanish is not sufficiently proficient for clinical assessment, and participation in a web-based educational program.
3. Participants who do not have sufficient vision and hearing to participate in an online educational program
4. Individuals who do not have the technical ability to participate in an online educational program. Technical ability is defined as ability to operate a computer/tablet and gain internet access; ability to send and receive emails)
5. Total Score on the T-MoCA <18
6. Individuals who have an advanced degree (e.g. Master's, MD, PhD) in an area related to brain health will not be eligible to participate.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Feldman, MDCM FRCP(C), Study Director — Alzheimer's Disease Cooperative Study (ADCS); Sarah Banks, PhD, ABPP-CN, Principal Investigator — Alzheimer's Disease Cooperative Study (ADCS)
Locations (1):
- Alzheimer's Disease Cooperative Study (ADCS), La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostergren JE, Heeringa SG, Leon CFM, Connell CM, Roberts JS. The Influence of Psychosocial and Cognitive Factors on Perceived Threat of Alzheimer's Disease. Am J Alzheimers Dis Other Demen. 2017 Aug;32(5):289-299. doi: 10.1177/1533317517714552. Epub 2017 Jun 13. PMID 28605999
- [Background] 2020 Alzheimer's disease facts and figures. Alzheimers Dement. 2020 Mar 10. doi: 10.1002/alz.12068. Online ahead of print. PMID 32157811
- [Background] Hurd MD, Martorell P, Delavande A, Mullen KJ, Langa KM. Monetary costs of dementia in the United States. N Engl J Med. 2013 Apr 4;368(14):1326-34. doi: 10.1056/NEJMsa1204629. PMID 23550670
- [Background] Agency, C.o.S.D.H.a.H.S., The Alzheimer's Project Clinical Rountable. Alzheimer's disease and related dementias in San Diego county. 2018.
- [Background] Living, A.f.C., Profile of Older Americans. 2019.
- [Background] Network, U.E.R.R.I.o.A.L.s., Latinos and Alzheimer's Disease: New Numbers Behind the Crisis. 2016.
- [Background] Velasco-Mondragon E, Jimenez A, Palladino-Davis AG, Davis D, Escamilla-Cejudo JA. Hispanic health in the USA: a scoping review of the literature. Public Health Rev. 2016 Dec 7;37:31. doi: 10.1186/s40985-016-0043-2. eCollection 2016. PMID 29450072
- [Background] Cummings J, Lee G, Ritter A, Zhong K. Alzheimer's disease drug development pipeline: 2018. Alzheimers Dement (N Y). 2018 May 3;4:195-214. doi: 10.1016/j.trci.2018.03.009. eCollection 2018. PMID 29955663
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Background] Cummings J, Reiber C, Kumar P. The price of progress: Funding and financing Alzheimer's disease drug development. Alzheimers Dement (N Y). 2018 Jun 13;4:330-343. doi: 10.1016/j.trci.2018.04.008. eCollection 2018. PMID 30175227
- [Background] Pendlebury ST, Welch SJ, Cuthbertson FC, Mariz J, Mehta Z, Rothwell PM. Telephone assessment of cognition after transient ischemic attack and stroke: modified telephone interview of cognitive status and telephone Montreal Cognitive Assessment versus face-to-face Montreal Cognitive Assessment and neuropsychological battery. Stroke. 2013 Jan;44(1):227-9. doi: 10.1161/STROKEAHA.112.673384. Epub 2012 Nov 8. PMID 23138443
- [Background] Chen, G., S.M. Gully, and D. Eden, Validation of a new general self-efficacy scale. Organizational research methods, 2001. 4(1): p. 62-83.
- [Background] Metlife Foundation. What America Thinks - Metlife Foundation Alzheimer's Survey. Available at: https://www.metlife.com/content/dam/microsites/about/corporateprofile/ alzheimers-2011.pdf. 2011.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cognitively normal midlife and older-adult participants were eligible to participate in this single arm pilot study. A total of 20 participants were enrolled at University of California San Diego. Recruitment began in March 2022 and the last participant exited the study August 2022. One participant withdrew from the study early.
Period: Overall Study
Arm/Group | HALT-AD
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | HALT-AD
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 12
  Latin American | 5
  More than one race | 1
  Unknown or prefer not to answer | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
Gender Identity [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Educational Attainment [Count of Participants; unit: Participants]
  Some high school | 1
  GED | 1
  Technical school or community college | 1
  Some university | 2
  Undergraduate degree at university | 6
  Some graduate (post-undergraduate school) | 1
  Graduate degree at university | 8
Geographic Area [Count of Participants; unit: Participants]
  Urban | 15
  Suburban | 5
Marital Status [Count of Participants; unit: Participants]
  Single | 2
  Married | 10
  Domestic partnership | 2
  Divorced | 4
  Widowed | 2
Housing type [Count of Participants; unit: Participants]
  House or apartment/condominium that you own | 11
  Apartment/condominium or house that you rent | 9

OUTCOME MEASURES:

1. Primary Outcome: Users' Engagement With the HALT-AD Online Platform by Measuring the Total Amount of Time (in Minutes) Spent Per User on All Courses Combined
Description: User engagement with the HALT-AD online platform by measuring the average total amount of time (in minutes) spent per user on all courses combined
Time Frame: 4 months
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | HALT-AD
Number analyzed (Participants) | 19
minutes | 136 [48.5 to 244]

2. Primary Outcome: Users' Engagement With the HALT-AD Online Platform by Measuring the Percentage of Participants Who Completed All Courses.
Description: Users' engagement with the HALT-AD online platform by measuring the percentage of participants who completed all courses.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | HALT-AD
Number analyzed (Participants) | 19
Participants | 10

3. Secondary Outcome: Change From Baseline in Knowledge on the HALT-AD Knowledge Assessment Survey at 4 Months
Description: The HALT-AD knowledge assessment survey is developed based on the HALT-AD program content to assess general knowledge of dementia including risk factors, brain health and prevention. Possible scores range from 0 (all answers are incorrect) to 20 (all answers are correct), with higher scores indicating greater knowledge of dementia. Change = (4 months score - baseline score). The greater the change in score, the greater the increase in knowledge of dementia.
Time Frame: at baseline and 4 months
Population: 14 out of 19 participants had completed the HALT-AD knowledge assessment survey at the end of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HALT-AD
Number analyzed (Participants) | 14
score on a scale | 1.18 (1.83)

4. Secondary Outcome: Change From Baseline in Self-efficacy on the New General Self-Efficacy Scale (NGSE) at 4 Months.
Description: The NGSE is an 8-item validated instrument assessing self-efficacy. Using a 5-point rating scale (1= strongly disagree to 5= strongly agree), participants report how much they believe they can achieve their goals. Total score for each participant is calculated by taking the mean of their ratings on each item, with the total possible score ranging from 1 to 5 and higher scores indicating greater self-efficacy. Change = (4 months score - baseline score). The greater the change in score, the greater the increase in self-efficacy.
Time Frame: at baseline and 4 months
Population: 14 out of 19 participants had completed the HALT-AD New General Self-Efficacy Scale (NGSE) survey at the end of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HALT-AD
Number analyzed (Participants) | 14
score on a scale | 0.1 (0.5)

5. Secondary Outcome: Change From Baseline in Lifestyle Risk on the HALT-AD Lifestyle Risk Assessment Survey at 4 Months
Description: The HALT-AD lifestyle risk assessment survey is developed by the HALT-AD subject- matter expert team to assess adherence to a potentially dementia risk-reducing lifestyle. Possible scores range from 3 (very high risk) to 15 (very low risk). Change = (4 months total score - baseline total score). The greater the change in score, the greater the increase in adherence to a potentially dementia risk-reducing lifestyle.
Time Frame: at baseline and 4 months
Population: 14 out of 19 participants completed the HALT-AD lifestyle risk assessment survey at the end of the study
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HALT-AD
Number analyzed (Participants) | 14
score on a scale | 1 [-0.75 to 1]

6. Other Pre Specified Outcome: Acceptability Survey- Users' Acceptability of the HALT-AD Program Content
Description: Qualitative evaluation of participant responses on the HALT-AD Course Acceptability Survey completed at 4 months
Time Frame: completed at 4 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: FOCUS Group Discussion- Qualitative Evaluation of the HALT-AD Program Content
Description: Qualitative evaluation of participant responses during the focus group discussion
Time Frame: 4 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Users' Satisfaction With the Facilitated Support Discussion Groups
Description: Qualitative evaluation of participant responses on the HALT-AD Facilitated Discussion Group Acceptability Survey
Time Frame: 4 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Qualitative Evaluation of Participant Responses During the Focus Group Discussion Groups
Description: Qualitative evaluation of participant responses during the focus group-discussion groups
Time Frame: 4 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Usability of the HALT-AD Program
Description: Users will complete the HALT-AD User Experience survey which is adapted for HALT-AD based on questions from the User Experience Questionnaire (UEQ) available at https://ueqtryitout.ueq-research.org/. Participants will be asked to decide as spontaneously as possible which conflicting terms (e.g. annoying vs. enjoyable) better describes the HALT-AD program. Additionally, users will complete the Net Promoter Score Survey (NPS) which asks one question "How likely is it that you would recommend HALT-AD to a friend or colleague?" and is reported on a scale of -100 (extremely unlikely) to +100 (extremely likely).
Time Frame: 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other(not including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (not including Serious) Adverse Events were not monitored/assessed.
Arm/Group | HALT-AD
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT05350410/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT05350410/ICF_001.pdf